CLINICAL TRIAL: NCT00807547
Title: A Randomised, Parallel-group, Double-blind, Placebo-controlled, Multicentre Phase III Trial Assessing the Pharmacodynamic Efficacy and Safety of an Intra-seasonal Short-time Updosing Schedule for Alutard SQ
Brief Title: Intraseasonal Short-time Up-dosing With Alutard SQ Grasses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHX0562
Record Dates: First submitted 2008-09-30; First posted 2008-12-12 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergy vaccination (Active Comparator): Allergy vaccination by 6 subcutaneous injections to 10,000 SQ-U with 1-3 days intervals, continuation by 2 injections with 10,000 SQ-U with 2-4 weeks intervals
  Interventions: Biological: Allergy vaccination (Alutard SQ)
- Subcutaneous injections (Placebo Comparator): Placebo injections
  Interventions: Biological: Allergy vaccination (Alutard SQ)

INTERVENTIONS:
Biological: Allergy vaccination (Alutard SQ) — Alutard SQ grasses and rye, 8 subcutaneous injections, updosing to 10.000 SQ-U, duration of treatment 50 days

SUMMARY:
Test of pharmacodynamic efficacy and tolerability of a short-time intra-seasonal updosing

ELIGIBILITY:
Inclusion Criteria:

* history of grass pollen induced allergic rhinoconjunctivitis
* positive skin prick test

Exclusion Criteria:

* uncontrolled severe bronchial asthma
* previous treatment with immunotherapy within the previous 5 years
* contraindication for specific immunotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Immuno globuline E (IgE)-blocking factor | 9 weeks

SECONDARY OUTCOMES:
Tolerability | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Klimek, MD, Principal Investigator — Center for Rhinology and Allergology, An den Quellen 10, 65183 Wiesbaden, Germany
Locations (1):
- Center for Rhinology and Allergology, Wiesbaden, Germany

REFERENCES:
- [Result] Pfaar O, Wolf H, Klimek L, Schnitker J, Wustenberg E. Immunologic effect and tolerability of intra-seasonal subcutaneous immunotherapy with an 8-day up-dosing schedule to 10,000 standardized quality-units: a double-blind, randomized, placebo-controlled trial. Clin Ther. 2012 Oct;34(10):2072-81. doi: 10.1016/j.clinthera.2012.09.006. PMID 23063373